CLINICAL TRIAL: NCT00396006
Title: The Effect of Augmentation Therapy With ARALAST Fraction IV-1 (ARALAST) Alpha1-Proteinase Inhibitor (α1-PI) on the Level of α1-PI and Other Analytes in the Bronchoalveolar (BAL) Epithelial Lining Fluid (ELF)
Brief Title: Efficacy and Safety Study of Augmentation Therapy With ARALAST Fraction IV-1 (Human Alpha 1 - Proteinase Inhibitor)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 460502
Record Dates: First submitted 2006-11-03; First posted 2006-11-06 (Estimated); Results first posted 2011-01-04 (Estimated); Last update posted 2021-05-13 (Actual); Status verified 2021-04

CONDITIONS: Alpha 1-Antitrypsin Deficiency
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency | interventions — alpha 1-Antitrypsin

INTERVENTIONS:
Biological: Alpha1-Proteinase Inhibitor — 60 mg/kg, weekly, intravenous infusion
  Other Names: ARALAST Fr.IV-1; ARALAST NP

SUMMARY:
The purpose of this study is to evaluate the effects of weekly augmentation therapy with ARALAST Fraction IV-1 (Fr IV-1) on epithelial lining fluid (ELF) alpha 1-proteinase inhibitor levels and other ELF analytes and to assess the safety of the treatment. Eligible subjects with a diagnosis of severe congenital alpha 1-antitrypsin deficiency will receive 8 consecutive weekly treatments with 60 mg/kg/week of functional ARALAST Fr IV-1 administered intravenously. The efficacy and safety assessments will include two bronchoscopies with bronchoalveolar lavage on study initiation and on study termination and multiple imaging and laboratory safety assessments. Each subject will participate for a minimum of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent.
* Male or female 18 years of age or older.
* Documented, endogenous serum α1-PI level < 40 mg/dL measured at screening (unless otherwise approved by the Sponsor) after a minimum of 28-day washout of any prior replacement therapy (if applicable).
* Phenotype Pi Z (which includes Pi*Z/Z, Pi*Z/Null, or Pi*Malton/Z), or Pi*Null/Null.
* Pulmonary functions at screening meeting the following criteria:

  1. Forced expiratory volume at 1 second (FEV1) >= 50% of predicted value; or
  2. FEV1 > 35% of predicted value and diffusing capacity for carbon monoxide > 45% of predicated value, with no supplemental oxygen therapy and < 3 pulmonary exacerbations or bronchitis requiring antibiotics/corticosteroids within the past 12 months).
* For any female of childbearing potential, a negative urine test for pregnancy within 7 days prior to the first bronchoalveolar lavage (BAL) visit and agreement to employ adequate birth control measures for the duration of the study.
* No clinically significant abnormalities detected on a 12-lead electrocardiogram (ECG) performed at the screening visit (ECG previously obtained within the past 12 months may be used, if available).
* Laboratory results obtained at the screening visit, meeting the following criteria:

  1. Serum alanine aminotransferase (ALT) <= 2 times upper limit of normal (ULN)
  2. Serum aspartate aminotransferase (AST) <= 2 times ULN
  3. Serum total bilirubin <= 2 times ULN
  4. Proteinuria < +2 on dipstick analysis
  5. Serum creatinine <= 1.5 times ULN
  6. Absolute neutrophil count (ANC) >= 1500 cells/mm3
  7. Hemoglobin (Hgb) >= 10.0 g/dL
  8. Platelet count >= 105/mm3
* If the subject is treated with respiratory medications, such as inhaled bronchodilators or inhaled corticosteroids, or other chronic medications for the treatment of the subjects´s other medical condition(s), the subject's medication doses were unchanged for at least 14 days prior to the baseline BAL visit.

Exclusion Criteria:

* Clinically significant pulmonary impairment, other than chronic pulmonary disease (COPD).
* The subject has received any alpha 1 proteinase inhibitor (α1-PI) augmentation therapy (e.g., Prolastin, Zemaira, Aralast, or an investigational α1-PI, by any route including intravenous and inhaled) within 28 days prior to screening.
* The subject has received an investigational drug or device within 1 month prior to screening, or the subject is currently receiving an investigational drug or device. If the subject receives another investigational drug or device after enrollment, the subjects is to be withdrawn from the trial.
* Presence of clinical symptoms of any lower respiratory tract infection or acute pulmonary exacerbation within 14 days prior to screening.
* The subject has a known selective Immunoglobulin A (IgA) deficiency (IgA level less than 15 mg/dL) and/or antibody against IgA.
* The subject is pregnant or lactating, or intends to become pregnant during the course of the study.
* The subject is not a suitable candidate for a BAL procedure.
* Moderate or severe bronchiectasis (total daily sputum production > 10 mL).
* Clinically significant medical, psychiatric, or cognitive illness, or recreational drug/alcohol use that, in the opinion of the investigator, would affect subject safety or compliance.
* Prior history of adverse reaction to local anaesthetics, sedatives, pain control drugs, and other medication employed at the study center for perioperative care associated with the BAL procedure.
* Long-term use of oral or parenteral glucocorticosteroid within 28 days prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-10-27 (Actual); Primary Completion 2007-12-14 (Actual); Study Completion 2007-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (5):
- Australia (3):
  - Adelaide, South Australia
  - Melbourne, Victoria
  - Nedlands, Western Australia
- New Zealand (2):
  - Otahuhu, Auckland
  - Hamilton

REFERENCES:
- [Derived] Li Z, Franke RM, Morris DN, Yel L. Pharmacokinetics and Biochemical Efficacy of an alpha1-Proteinase Inhibitor (Aralast NP) in alpha1-Antitrypsin Deficiency: a Cross-Product Retrospective Comparability Analysis. Pulm Ther. 2022 Sep;8(3):311-326. doi: 10.1007/s41030-022-00199-4. Epub 2022 Aug 24. PMID 36001294

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 5 hospital sites in New Zealand and Australia. The period studied was 1 year and 2 months.
Pre-assignment Details: 21 participants enrolled: 4 were screen failures (i.e., did not meet inclusion/exclusion criteria), 3 were discontinued due to unevaluable baseline bronchoalveolar lavage (BAL) samples, and 1 subject withdrew consent prior to receiving investigational product.
Groups:
- Participants Treated With ARALAST Fraction IV-1 (Fr. IV-1): Weekly infusions of ARALAST Fr. IV-1 were administered to participants at a dosage of 60 mg/kg
Period: Overall Study
Arm/Group | Participants Treated With ARALAST Fraction IV-1 (Fr. IV-1)
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Participants Treated With ARALAST Fr. IV-1
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 3
Age, Continuous [Median (Full Range); unit: years] | 59.6 [36.0 to 76.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 8
  New Zealand | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Bronchoalveolar Lavage (BAL) Epithelial Lining Fluid (ELF) Alpha1-Proteinase Inhibitor (α1-PI) Level
Description: Median change BAL ELF antigenic α1-PI level the from baseline to post-treatment
Time Frame: BAL procedures were performed at baseline and after 8 consecutive weeks of treatment (minimum of 12 weeks)
Population: Per protocol
Measure: Median (Full Range); unit: μM
Groups:
- Per Protocol: Treated participants with no major protocol violations, evaluable pre- and post-treatment BAL procedures, and 8 consecutive weekly treatments.
Arm/Group | Per Protocol
Number analyzed (Participants) | 10
μM | 0.28 [-0.24 to 4.90]
Statistical Analysis 1: Comparison: Per Protocol; Test type: Superiority or Other; p = 0.0195, Wilcoxon signed rank test

2. Primary Outcome: The Number of Adverse Events (AEs) Related to the Infusion of ARALAST Fr. IV 1 Administered at a Rate of 0.2 mL/kg/Min
Time Frame: During 8 consecutive weeks of treatment
Population: Intent to treat
Measure: Number; unit: adverse events
Groups:
- Intent to Treat: Treated participants with relevant assessments, e.g. if pre- and post-treatment BAL procedures were required to assess the parameter, then the participant had both evaluable BAL procedures.
Arm/Group | Intent to Treat
Number analyzed (Participants) | 13
adverse events | 0

3. Secondary Outcome: Ratio of Post- to Pre-treatment BAL ELF Antineutrophil Elastase Capacity (ANEC) Levels
Description: Median ratio of post- to pre-treatment BAL ELF ANEC levels
Time Frame: BAL procedures were performed at baseline and after 8 consecutive weeks of treatment (minimum of 12 weeks)
Population: Per protocol
Measure: Median (Full Range); unit: μM
Arm/Group | Per Protocol
Number analyzed (Participants) | 2
μM | 1.22 [0.63 to 1.81]

4. Secondary Outcome: Change in in the Ratio of BAL ELF α1-PI to Human Neutrophil Elastase (HNE) Complex Concentration
Description: Median change in the ratio of BAL ELF α1-PI to HNE complex concentration from baseline to post-treatment
Time Frame: BAL procedures were performed at baseline and after 8 consecutive weeks of treatment (minimum of 12 weeks)
Population: No per protocol subject had both pre- and post-treatment analytes available, therefore no analysis could be performed on this outcome measure
Arm/Group | Per Protocol
Number analyzed (Participants) | 0

5. Secondary Outcome: Change in the α1-PI Plasma Level
Description: Mean change in the plasma level of α1-PI from baseline to post-treatment
Time Frame: Blood samples were collected at baseline and after 8 consecutive weeks of treatment
Population: Per protocol
Measure: Mean (Standard Deviation); unit: μM
Arm/Group | Per Protocol
Number analyzed (Participants) | 12
μM | 10.34 (2.50)
Statistical Analysis 1: Comparison: Per Protocol; Test type: Superiority or Other; p < 0.0001, paired t-tests

6. Secondary Outcome: Change in the Plasma Antineutrophil Elastase Capacity (ANEC) Level
Description: Mean change in the plasma ANEC level from baseline to post-treatment
Time Frame: Blood samples were collected at baseline and after 8 consecutive weeks of treatment
Population: Per protocol
Measure: Mean (Standard Deviation); unit: μM
Arm/Group | Per Protocol
Number analyzed (Participants) | 12
μM | 9.46 (2.31)
Statistical Analysis 1: Comparison: Per Protocol; Test type: Superiority or Other; p < 0.0001, paired t-tests

7. Other Pre Specified Outcome: Change in the BAL ELF Free Neutrophil Elastase Level
Description: Median change in the BAL ELF Free Neutrophil Elastase Level from baseline to post-treatment
Time Frame: BAL procedures were performed at baseline and after 8 consecutive weeks of treatment (minimum of 12 weeks)
Population: Per protocol population with both pre- and post-treatment analytes available from BAL procedures
Measure: Median (Full Range); unit: nM
Arm/Group | Per Protocol
Number analyzed (Participants) | 3
nM | 41.17 [3.91 to 41.61]

8. Other Pre Specified Outcome: Ratio of Post- to Pre-treatment BAL ELF Total Neutrophil Elastase Level
Description: Median ratio of post- to pre-treatment BAL ELF Total Neutrophil Elastase Level
Time Frame: BAL procedures were performed at baseline and after 8 consecutive weeks of treatment (minimum of 12 weeks)
Population: Per protocol
Measure: Median (Full Range); unit: nM
Arm/Group | Per Protocol
Number analyzed (Participants) | 5
nM | 1.24 [0.47 to 30.97]
Statistical Analysis 1: Comparison: Per Protocol; Test type: Superiority or Other; p = 0.1875, Wilcoxon signed rank test

9. Other Pre Specified Outcome: Ratio of Post- to Pre-treatment BAL ELF Interleukin 8 (IL-8) Level
Description: Median ratio of post- to pre-treatment BAL ELF IL-8 Level
Time Frame: BAL procedures were performed at baseline and after 8 consecutive weeks of treatment (minimum of 12 weeks)
Population: Per protocol
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Per Protocol
Number analyzed (Participants) | 6
pg/mL | 1.46 [0.48 to 10.38]
Statistical Analysis 1: Comparison: Per Protocol; Test type: Superiority or Other; p = 0.4375, Wilcoxon signed rank

10. Other Pre Specified Outcome: Change in the BAL ELF Tumor Necrosis Factor-alpha (TNF-α) From Baseline to Post-treatment
Description: Median change in the BAL ELF TNF-α from baseline to post-treatment
Time Frame: BAL procedures were performed at baseline and after 8 consecutive weeks of treatment (minimum of 12 weeks)
Population: Per protocol population with both pre- and post-treatment analytes available from BAL procedures
Arm/Group | Per Protocol
Number analyzed (Participants) | 0

11. Primary Outcome: Number of Changes in the Rate of Infusion
Description: Number of decreases in the rate or discontinuations of infusion at 0.2 mL/kg/min
Time Frame: During 8 consecutive weeks of treatment
Measure: Number; unit: infusions
Arm/Group | Intent to Treat
Number analyzed (Participants) | 13
infusions | 0

12. Secondary Outcome: Clinically Significant Changes in Vital Signs From Pre- to Post-Infusion
Description: Clinically significant changes in vital signs from pre- to post-infusion are: • Heart rate: 25% increase above pre-infusion value • Blood pressure: ≥ 30 mm Hg change from pre-infusion blood pressure (systolic or diastolic) • Temperature: an increase in body temperature to >38°C (>100.4°F). If the pre-infusion body temperature was already >38°C (>100.4°F), then any further increase in body temperature by 1.1°C (1.98°F) or more was considered clinically significant. • Respiratory rate: 25% increase above pre-infusion value
Time Frame: During 8 consecutive weeks of infusion
Population: Intention to treat
Measure: Number; unit: # Clinically significant events
Arm/Group | Intent to Treat
Number analyzed (Participants) | 13
# Clinically significant events | 2

ADVERSE EVENTS:
Time Frame: 1 year, 2 months
Arm/Group | Intent to Treat
Serious Adverse Events (participants affected / at risk) | 1/13
Other Adverse Events (participants affected / at risk) | 7/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intent to Treat (N=13)
Hepatitis A antibody positive (Investigations) | 1 (1) — Not related to investigational product. This participant had received 2 Hepatitis A vaccinations in the year prior to enrollment.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intent to Treat (N=13)
Inflammation (General disorders) | 1 (1) — Not related to study drug
Sluggishness (General disorders) | 2 (2)
Vessel puncture site haematoma (General disorders) | 1 (1) — Not related to study drug
Bronchitis (Infections and infestations) | 1 (1) — Not related to study drug
Sinusitis (Infections and infestations) | 1 (1) — Not related to study drug
Contusion (Injury, poisoning and procedural complications) | 1 (1) — Not related to study drug
Post procedural complication (Injury, poisoning and procedural complications) | 2 (3) — Not related to study drug
Blood pressure systolic abnormal (Investigations) | 1 (1) — Not related to study drug
Respiratory rate increased (Investigations) | 1 (1) — Not related to study drug
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to study drug
Migrane (Nervous system disorders) | 1 (1)
Chest discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Not related to study drug
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (6)

LIMITATIONS AND CAVEATS:
Isoelectric focusing (IEF) analyses that were intended to compare the profile of plasma α1-PI & ELF α1-PI were not carried out due to fact that ELF samples were either missing, insufficient or too dilute for such assays.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The data from the study shall be published (if applicable) by the sponsor. The investigators and the steering committee may be involved if agreed to by the sponsor. Neither the investigator nor any other person within his/her institution has the right to publish separately or individually without permission by the sponsor.